CLINICAL TRIAL: NCT02881138
Title: A Phase I Study to Evaluate the Safety,Tolerability and Pharmacokinetics of RC48-ADC for Injection in Subjects With Advanced Malignant Solid Tumors With HER2-positive
Brief Title: A Study of RC48-ADC in Subjects With HER2-Positive Advanced Malignant Solid Tumors
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: RemeGen Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: C001 CANCER
Record Dates: First submitted 2016-08-20; First posted 2016-08-26 (Estimated); Last update posted 2020-07-30 (Actual); Status verified 2020-02

CONDITIONS: Solid Tumors

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- RC48-ADC (Experimental): Participants will be allocated to one of the following dose groups: 0.5, 1.0, 1.5, 2.0 and 2.5 mg/kg, and receive a treatment of RC48-ADC followed by 28 days of dose limited toxicity (DLT) observation period.
  Interventions: Drug: RC48-ADC

INTERVENTIONS:
Drug: RC48-ADC

SUMMARY:
A Phase I Study to Evaluate the Safety,Tolerability and Pharmacokinetics of RC48-ADC for Injection in Subjects With Advanced Malignant Solid Tumors With HER2-positive

ELIGIBILITY:
Inclusion Criteria:

* Signed informed consent form;
* Aged 18-65 years;
* ECOG physical condition is 0 or 1;
* Life expectancy greater than 12 weeks;
* Diagnosed with histologically or cytologically-confirmed, standard treatment is ineffective (disease progresses after treatment) or HER2-positive, locally advanced or metastatic malignant solid tumor patients who cannot tolerate standard therapy, cannot receive or do not have standard therapy;
* Human epidermal growth factor receptor 2 (HER2)-positive as measured either by immunohistochemistry (IHC 2+ and by fluorescence in situ hybridization (FISH) or by immunohistochemistry (3+);
* Patients with measurable and appreciable tumor lesions according to Response Evaluation Criteria in Solid Tumors (RECIST 1.1);
* Adequate organ function as defined by the following criteria:

  * absolute neutrophil count(ANC) >= 1.5 x 10(9)/L;
  * platelets>=100*10(9)/L;
  * Total serum bilirubin <=1.5*ULN;
  * serum aspartate transaminase (AST) and serum alanine transaminase (ALT) <=2.5*upper limit of normal (ULN), or AST and ALT<=5*ULN with hepatic metastasis;
  * Serum creatinine clearance rate >=45ml/min;
  * international normalized ratio (INR) and activated partial thromboplastin time (APTT) must be less than or equal to 1.5 times the upper limit of the normal range (ULN);
* Women of child-bearing potential and men must agree to use adequate contraception (e.g. condoms, implants, injectables, combined oral contraceptives, some intrauterine devices [IUDs], complete sexual abstinence, or sterilized partner) prior to study entry and during the period of therapy and for 30 days after the last dose of study drug;
* Left ventricular ejection fraction (LVEF) >= 50%.

Exclusion Criteria:

* Current pregnancy or lactation;
* Received anti-tumor treatment 4 weeks before study administration, including chemotherapy, radiotherapy, hormone therapy, biological therapy or immunotherapy, except the following: Gonadotropin-releasing hormone (GnRH) antagonistic therapy for prostate cancer and Hormone replacement therapy;
* Major surgery within 4 weeks of first dose of study drug and not fully recovered;
* Receiving palliative radiation therapy for bone metastases if administered <= 2 weeks prior to first study treatment;
* Toxicity of previous anti-tumor treatment has not recovered to CTCAE [version 4.0] 0-1 (with exception of alopecia);
* Participated in other clinical drug studies within 4 weeks;
* Hypersensitivity or delayed allergic reaction to certain components of RC48-ADC or similar drugs;
* According to the judgment of the investigator, a clinically significant active infection;
* A history of immunodeficiency, including a positive HIV test, or other acquired, congenital immunodeficiency diseases, or a history of organ transplantation;
* Uncontrollable systemic diseases including diabetes, hypertension, lung Fibrosis, acute lung disease, interstitial lung disease, etc.;
* Congestive heart failure with grade 2 or higher (including grade 2) by the New York Institute of Cardiology (NYHA) of the United States in the history of diseases such as acute myocardial infarction, unstable angina, stroke, or transient ischemic attack within 6 months before enrollment;
* Insufficient adherence to participate in this clinical study;
* Treated with Herceptin (Trastuzumab) within 60 days before the trial;
* Have received systemic steroid therapy for a long time ( short-term users who discontinue medication> 2 weeks can be selected);
* Uncontrolled primary or metastatic tumor of brain;
* Peripheral neuropathy with grade>= 2;
* People with a history of mental illness that is difficult to control.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2016-03-01 (Actual); Primary Completion 2020-04-30 (Actual); Study Completion 2020-07-15 (Actual)

PRIMARY OUTCOMES:
maximal tolerance dose (MTD) of RC48-ADC | DLT will be evaluated on 28 days of observation period
  Maximum-tolerated dose (MTD) was defined as the highest dose level at which no more than one of six patients experienced DLT during the DLT assessment window.
AEs | Estimated 2 years
  The drug safety was assessed by investigator(s) according to NCI-CTCAE v4.0

SECONDARY OUTCOMES:
Cmax | Estimated 2 years
  Maximum Observed Plasma Concentration
AUC | Estimated 2 years
  Area Under Curve
Tmax | Estimated 2 years
  Time for Cmax

CONTACTS AND LOCATIONS:
Overall Officials: Binghe Xu, Principal Investigator — Cancer Institute and Hospital, Chinese Academy of Medical Sciences
Locations (1):
- Cancer Hospital Chinese Academy of Medical Sciences, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided